CLINICAL TRIAL: NCT01425021
Title: Retrieval and Analysis of Orthopedic Implants at Revision Arthroplasty Surgery
Status: Completed | Type: Observational
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Christopher Peters, M.D., University of Utah
Other Study IDs: 43277
Record Dates: First submitted 2011-08-25; First posted 2011-08-29 (Estimated); Last update posted 2015-08-19 (Estimated); Status verified 2015-08

CONDITIONS: Total Joint Revisions

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Total hip/knee joint revisions: All University of Utah orthopedic patients who have had total or partial joint arthroplasties at the time of revision surgery.

SUMMARY:
The goal of this is to improve durability of total joint replacements in patients, thereby improving clinical outcomes and implant performance. To reach this objective, our research program would like to assess the safety, efficacy, performance, and durability of FDA approved biomaterial and implant designs used in joint replacements.

DETAILED DESCRIPTION:
The objective of the investigation will be to determine the mechanism of material failure and identify any design features that put the implant at risk for early failure. Normally all implants are discarded. The investigators will collect the implants indicated for removal and if there are impressive findings the investigators will perform research on the implants, otherwise the implants will be discarded. All patients will be followed prospectively after informed consent is signed. The implants that are chosen for research will be assessed for implant wear and failure at a lab appropriate for evaluating the particular concern.

ELIGIBILITY:
Inclusion Criteria:

* Patients who will be undergoing revision total joint surgery will be asked to participate in this study.

Exclusion Criteria:

* Patients who are not undergoing revision total joint surgery.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients undergoing revision total joint surgery.
Sampling Method: Non-Probability Sample
Enrollment: 199 (Actual)
Dates: Start 2010-08; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
determine the mechanism of material failure | 10 years

SECONDARY OUTCOMES:
identify any design features that put the implant at risk for early failure. | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Chris Peters, MD, Principal Investigator — University of Utah
Locations (1):
- University of Utah Orthopaedic Center, Salt Lake City, Utah, United States